CLINICAL TRIAL: NCT03134573
Title: PROmyBETAapp: Ascertaining Medication Usage & Documentation of Patient Reported Outcomes Utilizing the myBETAapp® in Patients With Multiple Sclerosis Treated With Betaferon®: a Pilot Study
Brief Title: Medication Usage and Patient Reported Outcomes Evaluation Via myBETAapp in Patients With Multiple Sclerosis Treated With Betaferon: a Pilot Study
Acronym: PROmyBETAapp
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 18462; BF1504 (Other: IMPACT)
Record Dates: First submitted 2017-04-26; First posted 2017-05-01 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Multiple Sclerosis
Keywords: Relapsing Remitting Multiple Sclerosis (RRMS),; Clinically isolated Syndrome (CIS),; Secondary Progressive Multiple Sclerosis (SPMS)
MeSH Terms: conditions — Multiple Sclerosis; Multiple Sclerosis, Relapsing-Remitting; Carcinoma in Situ; Multiple Sclerosis, Chronic Progressive | interventions — Interferon beta-1b

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Multiple Sclerosis: Women and men in Germany with the diagnosis of MS that are treated with Betaferon and use the myBETAapp
  Interventions: Drug: Interferon beta-1b (Betaferon, BAY86-5046); Device: Betaconnect auto-injector; Device: myBETAapp

INTERVENTIONS:
Drug: Interferon beta-1b (Betaferon, BAY86-5046) — Solution for injection
Device: Betaconnect auto-injector — Auto-injector for application of Betaferon solution which automatically covers injection related data
Device: myBETAapp — Medical device which can be connected with Betaconnect auto-injector and displays injection related data to patients and offers tracking of patient reported data at the wellness- tracker

SUMMARY:
The planned study will be a prospective, non-interventional, observational cohort study using the structure of a registry. Medication usage behavior will be observed for 6 months, while documentation behavior on the wellness tracker in the myBETAapp will be observed for 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 18 years.
* Patients on treatment with Betaferon (every Betaferon box contains a "Mixject" number, which is a product specific number unrelated to the study. Only patients prescribed Betaferon for their MS will be able to use the myBETAapp and participate in the study).
* Patients must be using the myBETAapp.
* Electronic informed consent must be obtained.

Exclusion Criteria:

-There are no exclusion criteria for participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of patients with multiple sclerosis who are treated with Betaferon and who are using the myBETAapp.
Sampling Method: Non-Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2017-09-15 (Actual); Primary Completion 2018-05-09 (Actual); Study Completion 2018-05-09 (Actual)

PRIMARY OUTCOMES:
Compliance to therapy (%) | 6 months
  Compliance (%) = ((true # of treatment days as derived from the data stored in the BETACONNECT)/(expected # of treatment days during observation period based on the injection frequency stipulated by the label))x100
Persistence of therapy (yes, no) | 6 months
  Persistence will be evaluated from the day of the first injection recorded in the BETACONNECT until the day of the last recorded injection or the end of observation (whichever comes first)
Adherence to therapy (yes, no) | 6 months
  Patients will be defined as being adherent to therapy if they fulfill the following criteria:
  1. They have been at least 80% compliant, i.e. applied ≥80% of the expected Betaferon injections and
  2. They have not dropped out of the study prior to the time of evaluation (i.e. they did not (1) stop using the myBETAapp or (2) withdraw their consent to participate in the study)

SECONDARY OUTCOMES:
Proportion of patients consenting to participate in this study among those using the myBETAapp | 3 months
  All patients registering their myBETAapp will be asked to participate in the study. Patients consenting to participate in the study will be flagged in the database. The proportion of patients consenting will then be calculated by dividing the number of patients giving consent by all patients asked.
Proportion of patients volunteering to record wellness related data in each of the following categories on the "Wellness chart" on the myBETAapp | 3 months
  Wellness Chart:(1) ability to walk, (2) coordination, (3) energy level, (4) bladder control, (5) exercise level,(6) memory, (7) vision, (8) bowel control, (9) emotions, and (10) eating habits

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many locations, Multiple Locations, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Limmroth V, Hechenbichler K, Muller C, Schurks M. Assessment of Medication Adherence Using a Medical App Among Patients With Multiple Sclerosis Treated With Interferon Beta-1b: Pilot Digital Observational Study (PROmyBETAapp). J Med Internet Res. 2019 Jul 29;21(7):e14373. doi: 10.2196/14373. PMID 31359863